CLINICAL TRIAL: NCT05768347
Title: Phase 1 Clinical Trial of Intravesical Adoptive Cell Therapy {ACT) With Tumor Infiltrating Lymphocytes (TIL) for Patients With BCG Exposed High Grade Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Intravesical Adoptive Cell Therapy w/ TIL for BCG Exposed High Grade NMIBC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21894
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma; Non-Invasive Bladder Urothelial Carcinoma
Keywords: Bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Adoptive Cell Therapy (Experimental): TIL from bladder biopsies will be propagated and cultured with interleukin-2 (IL-2) to a target goal of >30 million cells. These TIL then undergo rapid clonal expansion (REP) by incubation with anti-CD3 monoclonal antibody (mAb), resulting in >500-fold expansion. After 4-6 weeks culture time intravesical TIL will be administered via intravesical infusion, consisting of up to 3.2e8 cells in 40 mL aliquot. Intravesical therapy will be administered for up to 2 hours. This treatment will occur four times (Day 0, Day 7, Day 14 and Day 21).
  Interventions: Biological: Adoptive Cell Therapy with Tumor-infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Adoptive Cell Therapy with Tumor-infiltrating Lymphocytes (TIL) — Tissue samples are harvested, prepared and cryopreserved from post Bacillus Calmette-Guerin (BCG) bladder biopsies.

SUMMARY:
The purpose of the study is to evaluate the feasibility, safety and tolerability of intravesical adoptive cell therapy using TIL (tumor infiltrating lymphocytes) in participants with urothelial cell carcinoma (UCC) non-muscle invasive bladder cancer (NMIBC).

ELIGIBILITY:
Screening Inclusion Criteria:

* Bacillus Calmette-Guerin (BCG) exposed High Grade Non-Muscle Invasive Bladder Cancer (NMIBC) and healthy enough to participate:
* Histologically confirmed urothelial cell NMIBC (T1, Ta, and/or Tis) and: (a) bladder tumors with variant histology or mixed histology can be enrolled if the urothelial component is greater than 50% of the transurethral resection specimen (b) if Ta and T1, patients must have undergone complete restaging TURBT to confirm absence of muscle invasion (T2), however residual carcinoma in situ is acceptable. This restaging can be considered the primary tumor harvest if patients have had a previous resection.
* Have cytoscopic evidence of measurable disease. (There is no minimum measurement to be considered measurable disease. Any visible evidence is considered recurrence.)
* A tissue specimen may be obtained which is appropriate for TIL preparation. The tissue may be collected through a procedure the patient otherwise requires for treatment purposes. Alternatively, and in consultation with a surgical specialist, a separate procedure of limited risk to the patient (such as a repeat bladder biopsy) may be performed specifically for tissue collection purposes.
* ECOG performance status 0-1
* Participants must have adequate organ and marrow function in an assessment performed within 7 days (+ 3 day window) of enrollment as defined in protocol.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any previous treatment with intravesical chemotherapy within the previous 6 months.
* Current or prior use of any immunosuppressive medications, such as corticosteroids, within 14 days before enrollment. (a) Oral hydrocortisone, only for the purposes of a documented and confirmed adrenal insufficiency diagnosis, is permitted if ≤ 25 mg daily total dose. (b) Inhaled, intranasal, or topical corticosteroids are permitted.
* Current or prior use of anticancer therapy that has been shown to effect lymphocyte function before TIL collection.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than stable atrial fibrillation).
* Patients known to be HIV positive, hepatitis B or C positive, or both rapid plasma reagin (RPR) and fluorescent treponemal antibody (FTA) positive. (Hepatitis B surface or core antibody alone is not indicative of Hepatitis B Virus (HBV) infection).
* Known history of previous tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to first anticipated dose of TIL.
* History of allogeneic organ transplant
* History of primary immunodeficiency
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Patients with active systemic infections requiring intravenous antibiotics within 1 week prior to enrollment.
* Any unresolved toxicity (>CTCAE v5 grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy).
* History of pneumonitis or drug-related inflammatory lung disease.
* Active or prior documented autoimmune disease within the past 2 years. Note: Subjects with vitiligo, Grave's disease, limited site eczema, or limited site plaque psoriasis not requiring systemic treatment (within the past 2 years), or other autoimmune conditions which are not expected to recur, are allowed after approval from the medical monitor or PI.
* Patients with other prior malignancies must have had a ≥ 2-year disease-free interval, except for: in situ carcinoma of the cervix, in situ ductal carcinoma of the breast, in situ prostate cancer, in situ bladder cancer. These must have been deemed stable and not expected to relapse. In addition, early stage skin cancers, including basal, squamous cell cutaneous carcinoma, and melanoma, are permitted if previously treated with curative intent and not expected to relapse.
* Women who are pregnant or lactating.
* The effects of adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TIL) infusion on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and until 4 months after completion of study drug administration. Those who do not agree must be excluded. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. WOCBP are defined as premenopausal women capable of becoming pregnant.
* Penicillin allergy (Penicillin is used in the manufacturing of the cellular therapy product and therefore patients with a documented penicillin allergy are excluded from the trial)Patients with antibiotic allergies per se are not excluded; although the production of TIL for adoptive transfer includes antibiotics, extensive washing after harvest will minimize systemic exposure to antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Adoptive Cell Therapy with TILs | Up to 6 months
  Toxicity will be measured according to CTCAE v5. Investigators will determine if the serious toxicity rate exceeds 17%.

SECONDARY OUTCOMES:
Overall Response Rate | at 3 months
  Overall response is defined as the patient being alive 4 weeks after the adoptive TIL transfer, and the tumor size evaluated using the RECIST 1.1 criteria is consistent with a complete response (CR) or partial response (PR). The overall response (CR+PR) rate will be summarized using both a point estimate and its exact 95% confidence interval based on the binomial distribution.
Progression Free Survival | up to 12 months
  Progression-free survival (PFS), defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve. Confidence intervals for the median and survival rates at different time points will be constructed if needed and appropriate. This secondary endpoint will be reported descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Poch, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States